CLINICAL TRIAL: NCT01309490
Title: An Open-label, Dose Escalation Phase I/II Study of Ribavirin Given as Monotherapy in Solid Tumour Cancer Patients Expressing Elevated eIF4E
Brief Title: Phase I/II Study of Ribavirin Given as Monotherapy in Solid Tumour Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual, competing studies
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Wilson Miller, Professor - Department of Medicine, Division of Experimental Medicine, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ribavirin-004
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Malignant Solid Tumor
Keywords: high eIF4E expression; solid tumor cancer
MeSH Terms: interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ribavirin, nucleoside analog (Experimental)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — Dose Level: 1 1400 mg po BID Dose Level: 2 1800 mg po BID Dose Level: 3 2200 mg po BID Dose Level: 4 2600 mg po BID Dose Level: 5 3000 mg po BID

SUMMARY:
The purpose of this study is to learn whether oral Ribavirin is safe and effective in treating patients with solid tumour cancers, that have high levels of the protein eIF4E.

DETAILED DESCRIPTION:
This is a dose escalating, open-label, Phase I/II study of single agent oral ribavirin administered daily in solid tumour cancer patients who have failed standard treatments, overexpress eIF4E, and have easily accessible disease for serial biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I part of study : Histologically or cytologically confirmed cancer at diagnosis, with advanced, incurable disease at the time of screening, who have progressed on or are not suitable for standard therapy.

   Phase II part of study: Histologically or cytologically confirmed BC or HNSCC at diagnosis, with advanced, incurable disease at the time of screening, who have progressed on or are not suitable for standard therapy.
2. Willing to have a screening biopsy performed from an easily accessible lesion (ex. skin, superficial lymph node) AND whose tumour must overexpress eIF4E.
3. Easily accessible lesion for serial biopsies (ex. skin, superficial lymph node, or other easily accessible site).
4. At least 1 unidimensionally measurable lesion (based on the RECIST criteria) outside the CNS.
5. ECOG 0, 1, or 2.
6. Adequate recovery (excluding alopecia) from previous surgery, radiation, and chemotherapy.
7. Adequate wash-out period from last therapy (at least 3 weeks).
8. Life expectancy ≥ 12 weeks.
9. Age ≥ 18 years old.
10. Female patients of childbearing potential must have a negative serum (beta-HCG) pregnancy test within 14 days of starting protocol and must not be breastfeeding. Men and women of childbearing potential (including men who have had a vasectomy and women who have had tubal ligation) must agree to use two effective means of contraception throughout the study and for at least 6 months after completion of protocol. Post-menopausal women (defined as 12 or more consecutive months of amenorrhea, or follicle stimulating hormone (FSH) in the post-menopausal range), or surgically sterile women (defined as removal of the uterus or ovaries), do not require methods of contraception.
11. Adequate renal and hepatic function: serum creatinine < 1.5 x ULN; AST or ALT < 2.5 x ULN (or < 5 x ULN if liver involvement with metastases); serum bilirubin < 1.5 x ULN.
12. Adequate hematopoietic function: neutrophils ≥ 1.0 x 109/L, platelets ≥ 75 x 109/L.
13. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
14. Accessible for treatment and follow up.

Exclusion Criteria:

1. Symptomatic brain metastases.
2. Active cardiovascular disease as defined by New York Heart Association (NYHA) class III-IV categorization.
3. Intercurrent illness or medical condition precluding safe administration of the planned protocol treatment or required follow-up.
4. Use of any investigational anti-cancer drug within 2 weeks before start of study treatment or inadequate recovery from any toxic effects of such therapy.
5. Female patients who are pregnant or breastfeeding.
6. Concurrent treatment with other anti-cancer therapy. Bisphosphonates are allowed as long as they were started prior to screening (at least 4 weeks before study entry).
7. Known infection with HIV.
8. History of other malignancy in the past 5 years. Subjects who have been disease-free for 1 year or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03-17 (Actual); Primary Completion 2014-10-29 (Actual); Study Completion 2014-10-29 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) and/or recommended phase II dose (RP2D) | Average 1.5 years
Phase II: Determine the overall response rate to therapy with ribavirin | Average 1.5 years

SECONDARY OUTCOMES:
Incidence and nature of DLTs | 3 years
Incidence, nature and severity of adverse events | 3 years
Time to and duration of response, defined as the first occurence of documented objective response until the time of recurrence or death from any cause | 3 years
Clinical benefit rate, defined as the overall response rate and stable disease for greater than or equal to 24 weeks | 3 years
Pharmacokinetic parameters of ribavirin determine by total exposure, maximum plasma concentration, etc. | 3 years
Correlation between eIF4E activity and response | 3 years
To determine the effect of ribavirin on the activity of eIF4E related pathways through correlative studies | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Assouline S, Culjkovic B, Cocolakis E, Rousseau C, Beslu N, Amri A, Caplan S, Leber B, Roy DC, Miller WH Jr, Borden KL. Molecular targeting of the oncogene eIF4E in acute myeloid leukemia (AML): a proof-of-principle clinical trial with ribavirin. Blood. 2009 Jul 9;114(2):257-60. doi: 10.1182/blood-2009-02-205153. Epub 2009 May 11. PMID 19433856
- [Background] Kentsis A, Topisirovic I, Culjkovic B, Shao L, Borden KL. Ribavirin suppresses eIF4E-mediated oncogenic transformation by physical mimicry of the 7-methyl guanosine mRNA cap. Proc Natl Acad Sci U S A. 2004 Dec 28;101(52):18105-10. doi: 10.1073/pnas.0406927102. Epub 2004 Dec 15. PMID 15601771